CLINICAL TRIAL: NCT06398080
Title: Real-World Patient Characteristics, Treatment Patterns, and Outcomes Among Patients With Neovascular Age-Related Macular Degeneration (nAMD) and Diabetic Macular Edema (DME) Treated With Aflibercept 8 mg in the United States
Brief Title: An Observational Study to Investigate the Use of Aflibercept 8 mg to Treat Adult Patients With Neovascular Age-Related Macular Degeneration (nAMD) and Diabetic Macular Edema (DME) in a Real-World Setting
Acronym: SPECTRUM-US
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: VGFTe-HD-OD-2331
Record Dates: First submitted 2024-04-17; First posted 2024-05-03 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD); Wet Age-related Macular Degeneration (AMD); Diabetic Macular Edema (DME); Visual Impairment
Keywords: Treatment-Naïve; Previously treated; Degenerative disease; Vascular endothelial growth factor (VEGF); Diabetic retinopathy (DR)
MeSH Terms: conditions — Vision Disorders; Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Naïve nAMD: Treatment-naive patients with nAMD
  Interventions: Drug: aflibercept 8 mg
- Pretreated nAMD: Patients with nAMD who have been previously treated with anti-VEGF and/or laser
  Interventions: Drug: aflibercept 8 mg
- Naïve DME: Treatment-naive patients with DME
  Interventions: Drug: aflibercept 8 mg
- Pretreated DME: Patients with DME who have been previously treated with anti-VEGF, laser treatment, and/or intravitreal steroids
  Interventions: Drug: aflibercept 8 mg

INTERVENTIONS:
Drug: aflibercept 8 mg — No intervention will be provided to study patients. Any treatment decision, including the decision for aflibercept 8 mg treatment, is at the discretion of the attending physician, made in accordance with his/her experience and following approved clinical guidelines.
  Other Names: EYLEA® HD

SUMMARY:
The purpose of this research study is to observe the patient's clinical care and how EYLEA® HD is used as a treatment in real-world settings. Patients are asked to join the study because they have either neovascular age-related macular degeneration (nAMD/wet age-related macular degeneration [AMD]) or diabetic macular edema (DME). Patients cannot have used EYLEA® HD in the past and the doctor must be planning to treat nAMD or DME with a new prescription of EYLEA® HD (aflibercept 8 mg).

ELIGIBILITY:
Key Inclusion Criteria for Patients with nAMD:

1. Any patient aged at least 50 years at the time of enrollment
2. Diagnosis of nAMD (per physician)
3. Previously treated patient cohort, patients that had treatment with any ocular intervention for nAMD in the study eye at any time before starting aflibercept 8 mg, as defined in the protocol
4. For treatment-naïve patient cohort, patients never receiving previous treatment in the study eye for nAMD, as defined in the protocol
5. Initiating treatment with aflibercept 8 mg for nAMD

Key Inclusion Criteria for Patients with DME:

1. Any patient aged at least 18 years at the time of enrollment
2. Macular edema associated with DME (per physician)
3. Diagnosis of diabetes mellitus type 1 or type 2
4. For previously treated patient cohort, treatment with another intravitreal (IVT) anti-VEGF agent(s) or IVT steroids, or surgery/laser for DME in the study eye at any time before starting aflibercept 8 mg, as described in the protocol
5. For treatment-naïve patient cohort, patients never previously treated with IVT agents or surgery/laser in the study eye for DME
6. Initiating treatment with aflibercept 8 mg for DME

Key Exclusion Criteria for Patients with nAMD

1. Macular edema/hemorrhage/choroidal neovascularization due to any other cause besides nAMD
2. Any systemic or ocular condition that would prevent any improvement of VA in the study eye (eg, permanent visual impairment or blindness from any cause)
3. Any patients that have been treated with photodynamic therapy
4. Treatment with aflibercept 8 mg prior to baseline

Key Exclusion Criteria for Patients with DME:

1. Macular edema due to any other cause besides DME
2. Any systemic or ocular condition that would prevent any improvement of visual acuity in the study eye (eg, permanent visual impairment or blindness from any cause)
3. Treatment with aflibercept 8 mg prior to baseline

NOTE: Other Protocol-Defined Inclusion / Exclusion Criteria Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously treated and treatment-naïve patients that have a diagnosis of nAMD or DME will be enrolled into this study. Patients who are treated with aflibercept 8 mg for other indications besides nAMD or DME will not be included.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-12-12 (Estimated); Primary Completion 2028-01-03 (Estimated); Study Completion 2029-01-03 (Estimated)

PRIMARY OUTCOMES:
Mean prior treatment interval during the one-year period before study enrollment compared to the last assigned treatment interval during the study | Up to 12 Months
  Previously Treated Patient Cohorts:
  Reported among the subsets of patients (nAMD and DME) treated at dosing intervals of ≤ 8 weeks for ≥ 6 months prior to enrollment
Change in visual acuity (VA) (Early Treatment Diabetic Retinopathy study [ETDRS]) letters) | Baseline up to 12 Months
  Treatment-Naïve Patient Cohorts

SECONDARY OUTCOMES:
Change in VA (ETDRS letters) | Baseline up to 24 Months
Categorical gains of ≥5 ETDRS letters | Up to 24 Months
Categorical gains of ≥10 ETDRS letters | Up to 24 Months
Categorical gains of ≥15 ETDRS letters | Up to 24 Months
Categorical losses of ≥5 ETDRS letters | Up to 24 Months
Categorical losses of ≥10 ETDRS letters | Up to 24 Months
Categorical losses of ≥15 ETDRS letters | Up to 24 Months
Proportion of patients achieving 20/40 Snellen equivalent or better | Up to 24 Months
Change in Central subfield thickness (CST) | Baseline up to 24 Months
Description of demographics | At Baseline
  Standard and clinical characteristics such as age, sex and race/ethnicity
Descriptions of study eye characteristics | At Baseline
  Study eye characteristics include ocular history, medical history (duration of nAMD or DME), prior and concomitant medication history, prior and concomitant ocular surgeries
Treatment interval | Up to 24 Months
Missed and unscheduled visits | Up to 24 Months
Frequency of ocular adverse events (AEs) | Up to 24 Months
Frequency of non-ocular adverse events (AEs) | Up to 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals